CLINICAL TRIAL: NCT04341766
Title: Prospective Descriptive Study on the Evolution of Pulmonary Ultrasound in Patients Hospitalized for Covid19
Brief Title: Evolution of Pulmonary Ultrasound in Patients Hospitalized for Covid (Coronavirus Disease) 19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-ECHO
Record Dates: First submitted 2020-04-01; First posted 2020-04-10 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Pneumonia, Viral; COVID-19
MeSH Terms: conditions — Pneumonia, Viral; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient hospitalised with COVID-19 infection: Patients admitted to hospital with proven COVID-19 infection with respiratory signs warranting a chest CT scan
  Interventions: Other: No special intervention

INTERVENTIONS:
Other: No special intervention — No special intervention : Ultrasound data will be collected

SUMMARY:
Clinical thoracic ultrasound plays an important role in the exploration, diagnosis and follow-up of thoracic pathologies.

The COVID (Coronavirus Disease) epidemic is leading to a large influx of patients in the emergency department with respiratory disorders. The rapid diagnosis of respiratory disorders in infected patients is important for further management.

Chest ultrasound has already demonstrated its value in the diagnosis of pneumonia in the emergency department with superiority over chest X-ray.

However, there is little data on the thoracic ultrasound semiology of viral pneumonia in general and of COVID in particular.

DETAILED DESCRIPTION:
Chest ultrasound has already shown its value in the diagnosis of pneumonia in the emergency department with superiority over chest X-ray.

However, there is little data on the thoracic ultrasound semiology of viral pneumonia in general and of COVID in particular.

Peng reported data from 20 patients and compared them to chest CT. The abnormalities are a thickening of the pleuropneumonia line, an interstitial syndrome with B lines, corresponding to frosted glass opacities, confluent B lines (snowstorm appearance) corresponding to interstitial infiltrate, sub-pleural alveolar opacities corresponding to sub-pleural condensations, more frank alveolar images corresponding to alveolar opacities. A multifocal aspect was associated with involvement of more than 2 lobes. However, the frequency of these abnormalities as well as the sensitivity of the echo are not detailed in this article.

Another Italian article describes a clinical case of COVID-19 pneumonia with sub-pleural involvement and irregularity of the pleuro-pulmonary line.

Clinical thoracic ultrasound has a major potential interest during the COVID epidemic: available at the patient's bedside, avoiding the need to move around, feasible for the physician during his visit, easy to clean especially if ultraportable devices are used, fast and not exposing the staff any more than the usual clinical examination.

In order to determine whether this technique is useful in the management of infected patients or patients suspected of COVID-19 infection with respiratory signs, we propose a descriptive prospective study evaluating the ultrasound semiology of COVID-19 pneumonia and the interest of ultrasound in the evolutionary follow-up of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with proven COVID-19 infection with respiratory signs warranting a chest CT scan

Exclusion Criteria:

* Patient not agreeing to have his or her data collected for the study
* Unconscious patient

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to hospital with proven COVID-19 infection with respiratory signs and who need an hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Characteristics of pulmonary ultrasound for Covid-19 patients | Day one
  description of ultrasound abnormalities for Covid-19 patients

SECONDARY OUTCOMES:
Characteristics of pulmonary ultrasound for Covid-19 patients | Day 3
  description of ultrasound abnormalities for Covid-19 patients
Characteristics of pulmonary ultrasound for Covid-19 patients | Day 14
  description of ultrasound abnormalities for Covid-19 patients
Charateristics of pulmonary CT-scan for Covid-19 patients | Day 1
  description of CT-scan abnormalities for Covid-19 patients
Charateristics of pulmonary CT-scan for Covid-19 patients | Day 3
  description of CT-scan abnormalities for Covid-19 patients
Charateristics of pulmonary CT-scan for Covid-19 patients | Day 14
  description of CT-scan abnormalities for Covid-19 patients

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - CHU Amiens, Amiens
  - CH de la Côte Basque, Bayonne
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CHU Caen, Caen
  - CHG de Chambery, Chambéry
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU de Limoges, Limoges
  - APHM - Hopital Nord, Marseille
  - CHU de Nancy, Nancy
  - CHU Nîmes, Nîmes
  - CHR Orléans, Orléans
  - CHU Cochin, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen, Rouen
  - CH Saint-Quentin, Saint-Quentin
  - CHU Larrey - Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No